CLINICAL TRIAL: NCT01764919
Title: Exploration of the Use of [124I]FIAU Positron Emission Tomography-Computed Tomography Scanning in Diagnosing Osteomyelitis in Patients With Diabetic Foot Infection.
Brief Title: [124I]FIAU PET-CT Scanning in Diagnosing Osteomyelitis in Patients With Diabetic Foot Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No correlation between FIAU uptake and bone biopsy results.
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BVD003
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Foot Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [124I]FIAU (Experimental): Single intravenous injection of [124I]FIAU in patients with diabetic foot infection
  Interventions: Radiation: [124I]FIAU

INTERVENTIONS:
Radiation: [124I]FIAU — A single intravenous injection of 5 mCi[124I]FIAU in patients with diabetic foot infection who will undergo 2 PET-CT scanning.

SUMMARY:
This protocol will evaluate the sensitivity and specificity of [124I]FIAU as a diagnostic imaging agent for the detection of osteomyelitis in patients with diabetic foot infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients >/= 18 years on the day of signing consent.
2. A diagnosis of diabetes mellitus, type I or II, as evidenced either by HbA1c>6.5% or receipt of antidiabetic medication at time of enrollment.
3. Ability to provide informed consent
4. An inframalleolar ulcer of perfusion, extent/size, depth/tissue loss, infection and sensation (PEDIS) grade 2 or 3. At the discretion of the Investigator, patients with PEDIS grade 4 infections may be included if they are sufficiently stable.
5. For females of childbearing potential, a negative urine pregnancy test on the day of dosing.
6. For females of childbearing potential, a willingness to use 2 methods of contraception for 30 days after receiving [124I]FIAU.
7. Ability to return for all study assessments.
8. Clinically euthyroid, or on stable thyroid replacement therapy.

Exclusion Criteria:

1. Patients who ar unable to comply with study requirements.
2. Indication, in the opinion of the principal Investigator for urgent surgery that would preclude the time needed for PET-CT scanning, or clinical instability that precludes PET-CT scanning.
3. History of an inherited mitochondrial disorder (eg. Leber's hereditary neuropathy, neuropathy, ataxia, retinitis pigmentosa and ptosis [NARP], myoneurogenic gastrointestinal encephalopathy [MNGIE], myocolonic epilepsy with ragged red fibers [MERFF] and mitochondrial myopathy, encephalomyopathy, lactic acidosis and stroke-like syndrome [MELAS])
4. Alanine aminotransferase (ALT)>5x Upper Limit of Normal (ULN) OR aspartate aminotransferase (AST) >5x ULN.
5. Body mass that exceeds the rating of the CT table.
6. Hypersensitivity to iodine.
7. Pregnant or breast-feeding.
8. Any condition that would put the patient at unreasonable risk in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | [124I]FIAU
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Assess the Sensitivity and Specificity of [124I]FIAU PET-CT Scanning in Detecting Osteomyelitis as Determined by Bone Biopsy in Patients With Diabetic Foot Infection.
Description: A bone biopsy was obtained through a noninfected area and submitted for histology and microbiologic culture. Cultures were also to be obtained by biopsy after debridement of the ulcer from a clean base. Subjects were dosed with [124I]FIAU. PET-CT scanning were performed. All PET, PET-CT, and CT images, both attenuation corrected and uncorrected, were to be evaluated centrally and independently. Results from the bone biopsies were not available to the central reader of the PET-CT images. The sensitivity and specificity of [124I]FIAU PET-CT scanning in detecting osteomyelitis was determined based on its correlation with bone biopsy, the truth standard.
Time Frame: 30 hours
Measure: Number; unit: participants
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 4
participants
  Patient positive with both PET-CT and bone biopsy | 0
  Patient negative with both PET-CT and bone biopsy | 1
  Patient positive with PET-CT only | 1
  Patient positive with bone biopsy only | 2

2. Secondary Outcome: Assess the Safety and Tolerability of [124I]FIAU
Description: Safety will be monitored for all subjects for the duration of their study participation. Safety will be assessed by monitoring of adverse events,vital signs, physical exams, and clinical laboratory tests including CBC and serum chemistry.
Time Frame: 30 +/- 2 days
Measure: Number; unit: participants with adverse events
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 4
participants with adverse events | 2

3. Secondary Outcome: Compare the Sensitivity and Specificity of [124I]FIAU PET-CT Scanning to Gadolinium-enhanced (GE) Magnetic Resonance Imaging (MRI) and Non-GE-MRI Scanning in Detecting Osteomyelitis in Patients With Diabetic Foot Infection
Description: All PET-CT images will be evaluated centrally and independently by a single radiologist. Diagnosis of osteomyelitis based on PET-CT will be compared with MRI which is currently the test of choice to diagnose osteomyelitis in diabetic foot infection.
Time Frame: -2 to 72 hours post dose [124I]FIAU
Population: No correlation was seen between FIAU uptake and bone biopsy results (the standard of truth). The secondary and exploratory efficacy endpoints were not assessed.
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 0

4. Secondary Outcome: Assess Any Additional Information That [124I]FIAU PET-CT Scanning Provides Compared to MRI
Description: Additional information on the extent and localization of infection will be compared to MRI.
Time Frame: -2 to 72 hours post dose [124I]FIAU
Population: as for outcome 3
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Explore the Performance of [124I]FIAU PET-CT Compared to MRI in Detecting Osteomyelitis by Chronic Kidney Disease (CKD) Stage (Stage 1+2, Stage 3, and Stage 4+5).
Time Frame: -2 hours to 72 hours post dose [124I]FIAU
Population: as for outcome 3
Arm/Group | [124I]FIAU
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | [124I]FIAU
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [124I]FIAU (N=4)
wound dehiscence (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [124I]FIAU (N=4)
mild gamma-glutamyl transferase (GGT) increased (Investigations) | 1
anemia (Blood and lymphatic system disorders) | 1
nausea (Gastrointestinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
hypoglycemia (Blood and lymphatic system disorders) | 1
chronic renal failure (Renal and urinary disorders) | 1
mild blood alkaline phosphatase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days